CLINICAL TRIAL: NCT05105776
Title: Multimodal Neuromodulation in Individuals With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ryan D'Arcy (Industry)
Collaborators: Pacific Parkinson's Research Institute (Unknown); University of British Columbia (Other)
Responsible Party: Sponsor-Investigator, Ryan D'Arcy, Principal Investigator, HealthTech Connex Inc.
Organization: HealthTech Connex Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNS_PD_001
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Galvanic stimulation is masked (sham vs active)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physiotherapy only (No Intervention)
- Active galvanic stimulation (GVS; week 1) to sham GVS (week 2) (Experimental): Physiotherapy + translingual neurostimulation provided throughout
  Interventions: Device: Galvanic stimulation
- Sham GVS (week 1) to active GVS (week 2) (Experimental): Physiotherapy + translingual neurostimulation provided throughout
  Interventions: Device: Galvanic stimulation
- Active GVS throughout weeks 1 + 2 (Experimental): Physiotherapy + translingual neurostimulation provided throughout
  Interventions: Device: Galvanic stimulation

INTERVENTIONS:
Device: Galvanic stimulation — Galvanic stimulation during physiotherapy sessions
  Arms: Active GVS throughout weeks 1 + 2; Active galvanic stimulation (GVS; week 1) to sham GVS (week 2); Sham GVS (week 1) to active GVS (week 2)

SUMMARY:
Multimodal non-invasive neuromodulation paired with physical therapy is a promising treatment modality for Parkinson's Disease ("PD"), however the optimal stimulation method, dose, and associated therapeutic protocol for long-lasting clinical benefits have not yet been identified for this population.

Here the investigators aim to develop and execute a preliminary clinical study exploring the potential benefits of multimodal non-invasive neuromodulation. The therapeutic intervention will involve translingual neurostimulation +/- galvanic neurostimulation, paired with an intensive physical and cognitive therapy program.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of idiopathic PD
2. Disease staging between II and III (mild to moderate), according to the modified Hoehn and Yahr scale;
3. Currently taking prescribed antiparkinsonian medication regularly with:
4. No medication changes in the last 30 days
5. Responsive to oral dopamine replacement therapy
6. Score higher than 24, verified through the Montreal Cognitive Assessment33.
7. Must demonstrate moderate burden of motor symptoms (MDS-UPDRS part II >12 and MDS-UPDRS part III scores >35) 34
8. Must be able to voluntarily give written (or verbal) informed consent
9. Must have ability to reliably use the devices
10. Must be able to understand and complete all assessments (provided in English only)

    Exclusion Criteria:
11. Diagnosis of atypical parkinsonism;
12. History of epilepsy
13. Presence of an implanted electrical device
14. Previous surgical intervention for PD (DBS implantation - deep brain stimulation);
15. Treated with a pump for continuous delivery of DRT (Dopamine replacement therapy)
16. Presence of severe freezing episodes.
17. Women who are pregnant or nursing
18. History of unstable mood disorder or unstable anxiety disorder or psychosis
19. Those with a recent history of substance abuse and/or dependence (alcohol or other drugs)
20. Have been diagnosed with neurological disease other than Parkinson's disease.
21. Have a major concomitant illness or illnesses including cancer or disease of the cardiovascular, respiratory and/or renal systems deemed significant medical risk in the opinion of the principle investigator
22. Have a diagnosed vestibular dysfunction
23. Have had eye surgery within the previous three months or ear surgery within the previous six months
24. Have participated in another clinical trial within the last 30 days or are currently enrolled in another interventional clinical trial
25. Contraindicated for PoNS, including:

    25.1. Current disease or sensitivity of the oral cavity 25.2. History of oral cancer 25.3. Oral surgery within three months of screening 25.4. Oral cavity piercings that could interfere with PoNSTM use 25.5. Sensitivity to Nickel, Copper, or Gold 25.6. Currently enrolled in a PoNSTM treatment program or use of the PoNSTM device in the last 5 weeks 25.7. History of penetrating brain injuries 25.8. Chronic infectious disease 25.9. Unmanaged hypertension 25.10. Diabetes 25.11. History of seizures
26. Contraindicated for GVS, including:

26.1. Metallic brain implant(s) 26.2. Brain surgery within the past six months 26.3. Highly sensitive skin behind the ears

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
NeuroCom Sensory Organization Test (SOT) | Baseline to week 4
  Composite balance score
NeuroCom Limits of Stability test (LOS) | Baseline to week 4
  Postural stability score
NeuroCom Adaptation Test | Baseline to week 4
  Adaptation score
MiniBESTest | Baseline to week 4
  Balance score

SECONDARY OUTCOMES:
Electroencephalography - amplitudes | Baseline to week 4
  Measured with NeuroCatch Platform 2 (NCP)
Electroencephalography - latencies | Baseline to week 4
  Measured with NeuroCatch Platform 2 (NCP)
Unified Parkinson's Disease Rating Scale | Baseline to week 4
  Part II and part III: Motor function score
Montreal Cognitive Assessment (MoCA) | Baseline to week 4
  Cognitive test; total score

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Neurology Studies, Surrey, British Columbia, Canada